CLINICAL TRIAL: NCT05626504
Title: Outcome Study of the Pipeline Embolization Device With Vantage Technology in Unruptured Aneurysms
Acronym: PEDVU
Status: Active, not recruiting | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 317314
Record Dates: First submitted 2022-11-01; First posted 2022-11-23 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Brain Aneurysm; Intracranial Hemorrhages; Stroke
MeSH Terms: conditions — Intracranial Aneurysm; Intracranial Hemorrhages; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Pipeline Embolization Device with Vantage Technology — Flow-diverter device occludes aneurysms through endoluminal reconstruction and remodelling of the parent artery.

SUMMARY:
In this project the investigators study the safety and efficacy of the pipeline embolization device with vantage technology in treatment of unruptured brain aneurysms

ELIGIBILITY:
Inclusion Criteria:

* All patients treated with Pipeline Embolization Device with Vantage Technology (PEDV)
* MRA and/or DSA (or tomographic angiography) available for follow up

Exclusion Criteria:

* Insufficient background data available e.g., to determine size of aneurysm and pipeline device
* PEDV used for causes other than aneurysms, e.g., fistulas and dissection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Treated with pipeline embolization devices during 2021 and 2022
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-10-27 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate 30-day morbidity rates | Done at 30 days post procedural
  We will evaluate short term clinical outcome in the form of morbidity rates 30 days after the procedure
Evaluate 30-day mortality rates | Done at 30 days post procedural
  We will evaluate short term clinical outcome in the form of mortality rates 30 days after the procedure

SECONDARY OUTCOMES:
Evaluate 1-year morbidity rates | Done at >30days up to 1 year post procedural
  We will evaluate long term clinical outcome in the form of morbidity rates >30days up to 1 year after the procedure
Evaluate 1-year mortality rates | Done at >30days up to 1 year post procedural
  We will evaluate long term clinical outcome in the form of mortality rates >30days up to 1 year after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Kings College Hospital, London, United Kingdom

REFERENCES:
- [Background] Atasoy D, Kandasamy N, Hart J, Lynch J, Yang SH, Walsh D, Tolias C, Booth TC. Outcome Study of the Pipeline Embolization Device with Shield Technology in Unruptured Aneurysms (PEDSU). AJNR Am J Neuroradiol. 2019 Dec;40(12):2094-2101. doi: 10.3174/ajnr.A6314. Epub 2019 Nov 14. PMID 31727754